CLINICAL TRIAL: NCT03394794
Title: Study of the Efficacy of Treatment of Fecal Incontinence in Community-dwelling Women: Assessment of Individual Efficacy on Anorectal Physiology and Cortical Plasticity, Its Impact on Clinical Severity and on Quality of Life.
Brief Title: Study of the Efficacy of 4 Treatments for Fecal Incontinence in Community-dwelling Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Lluís Mundet, GI motility clinician / researcher, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IF02-11/2012
Record Dates: First submitted 2017-11-29; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Fecal Incontinence
Keywords: anorectal physiology; therapies; quality fo life
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kegel exercises (Active Comparator): Pelvic floor exercises designed in the 1950s' by Arnold Kegel.
  Interventions: Device: Pelvic floor rehabilitation
- biofeedback (Experimental): Biofeeback therapy to improve neuromuscular coordination and strengthen sphincter contractility.
  Interventions: Device: Pelvic floor rehabilitation
- electrostimulation (Experimental): Administration of electric current with a specific device (stimulator) and through a vaginal prove, in order to improve pelvic floor contractility.
  Interventions: Device: Pelvic floor rehabilitation
- transcutaneous neuromodulation (Experimental): Stimulation of tibial nerve with a specific electric current through a stimulator and surface electrodes
  Interventions: Device: Pelvic floor rehabilitation

INTERVENTIONS:
Device: Pelvic floor rehabilitation — The aim is to compare how each treatment improves symptoms and quality of life and which physiologic mechanisms affects. The basal treatment which other therapies are compared to is Kegel.

SUMMARY:
This is a RCT aimed to assessing efficacy of kegel exercises,biofeedback, electrostimulation and transcutaneous neuromodulation on women with fecal incontinence, measuring its impact on anorectal physiology, cortical plasticity, clmical severity and the quality of life.

DETAILED DESCRIPTION:
Fecal incontinence is a prevalent condition with a major impact on quality of life. Currently four treatments are being used in clinical practice: Kegel exercises (K), biofeedback (BF), electrostimulation (ES) and transcutaneous neuromodulation (NM). Results in the literature are discordant and lack methodological rigour making scientific evidence weak.

The aim of this study is to assess the efficacy of these four treatments on community-dwelling women and their impact on anorectal physiology, on clinical severity and on QoL.

This is a randomized control trial. Patient physiology was studied with anorectal manometry and endoanal ultrasonography; clinical severity was assessed with Cleveland and St. Mark's scales, and QoL with the Faecal Incontinence Quality of Life (FIQL) and the EuroQol's EQ5D questionnaires. Urinary incontinence (UI) was also evaluated by means of International Consultation on Incontinence (ICIQ) score. Patients were randomized and assigned to K (control), BF+K, ES+K or NM+K, given active treatment for a 3-month period, and then evaluated again with identical tests and parameters to identify changes.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18
* To be woman
* Have had incontinence episiodes at least from 6 month since the beginning of the study
* Have had incontinence episodes during the last month prior the beginning of the study
* The patient is able to understand the nature and impliations of the study and, therefore, to decide her participation.

Exclusion Criteria:

* Not meeting inclusion criteria
* Have very mild condition (Wexner <4)
* To be unable to perform / understand the treatments properly
* Being pregnant
* To have used treatmets for fecal incontinence within the last six months prior to the start of the study
* If, at reserarcher's criteria, the patient has not the proper conditions to perform and finish the treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
clinical severity | Changes of severity after 3 month-treatment
  severity of the symptoms measured with Cleveland score
maximum anal resting pressure | Changes maximum anal resting pressure after 3 month-treatment
  pressure of the anal canal measured with mmHg
maximum squeeze pressure | Changes maximum squeeze pressure after 3 month-treatment
  pressure on the anal canal when squeezing measured with mmHg
rectal sensitivity | changes in rectal balloon filling after 3 month-treatment
  patient's rectal perception, measured with cm3 of distention of a rectal balloon

IPD SHARING:
Plan to Share IPD: No